CLINICAL TRIAL: NCT00959231
Title: Transplantation of Umbilical Cord Blood From Unrelated Donors in Patients With Haematological Diseases Using a Reduced Intensity Conditioning Regimen
Brief Title: Donor Umbilical Cord Blood Transplant After Cyclophosphamide, Fludarabine Phosphate, and Total-Body Irradiation in Treating Patients With Hematologic Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cancer Research UK (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000643641; CRUK-UCL-RIC-UCBT; EUDRACT-2004-003845-41; EU-20946
Record Dates: First submitted 2009-08-13; First posted 2009-08-14 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2010-04

CONDITIONS: Hematopoietic/Lymphoid Cancer
Keywords: hematopoietic/lymphoid cancer
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Cyclophosphamide; Cyclosporine; fludarabine phosphate; Mycophenolic Acid; Cord Blood Stem Cell Transplantation; Whole-Body Irradiation

INTERVENTIONS:
Drug: cyclophosphamide
Drug: cyclosporine
Drug: fludarabine phosphate
Drug: mycophenolate mofetil
Other: laboratory biomarker analysis
Procedure: nonmyeloablative allogeneic hematopoietic stem cell transplantation
Procedure: umbilical cord blood transplantation
Radiation: total-body irradiation

SUMMARY:
RATIONALE: Giving low doses of chemotherapy and total-body irradiation before a donor umbilical cord blood transplant helps stop the growth of abnormal cells. It also stops the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune cells and help destroy any remaining abnormal cells (graft-versus-tumor effect). Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving cyclosporine and mycophenolate mofetil before and after transplant may stop this from happening.

PURPOSE: This phase II trial is studying the side effects of donor umbilical cord blood transplant after cyclophosphamide, fludarabine phosphate, and total-body irradiation in treating patients with hematologic disease.

DETAILED DESCRIPTION:
OBJECTIVES:

* To assess the safety and efficacy of unrelated-donor umbilical cord blood transplantation (UCBT) using a nonmyeloablative preparative regimen in patients with hematological disease, in a multi-institution UK setting.
* To confirm that unrelated-donor UCBT following nonmyeloablative conditioning is associated with consistent and durable engraftment in these patients.
* To assess transplant-related mortality at day 100 associated with nonmyeloablative UCBT in these patients.
* To assess the incidence of grades II-IV and III-IV acute graft-vs-host disease (GVHD) in these patients.
* To assess the risk of relapse and progressive disease in these patients at 1 year post transplant after nonmyeloablative UCBT.
* To assess overall and progression-free survival of these patients at 1 year after nonmyeloablative UCBT.
* To assess immune reconstitution at 1, 2, 3, 6, 12, and 24 months after transplant as measured by quantitative recovery of B, T, and NK cells (flow cytometry), qualitative recovery of T cells (TREC and spectratyping), in vivo functional T-cell responses (EBV and CMV tetramers), and quantitative immunoglobulins.

OUTLINE: This is a multicenter study.

* Reduced-intensity conditioning regimen: Patients receive cyclophosphamide IV over 2 hours on day -6 and fludarabine phosphate IV over 1 hour on days -6 to -2. Patients undergo a single fraction of total-body irradiation on day -1.
* Umbilical cord blood (UCB) transplantation: Patients undergo umbilical cord blood transplantation on day 0.
* Graft-vs-host disease prophylaxis: Patients receive cyclosporine IV or orally on days -3 to 100 followed by taper and mycophenolate mofetil IV or orally on days -3 to 35 followed by taper.

Blood and bone marrow samples are collected periodically for analysis.

After completion of study treatment, patients are followed up every 3 months in year 1, every 4 months in year 2, every 6 months until 5 years, and then annually thereafter.

Peer Reviewed and Funded or Endorsed by Cancer Research UK.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of high-risk, advanced or poorly responding hematological disease for which a reduced-intensity hemopoietic stem cell transplantation is likely to be effective

  * Disease status is such that there is no alternative therapy likely to achieve a cure or provide a significant prolongation of disease-free survival
* No chronic myelogenous leukemia in first chronic phase responding to imatinib or refractory blast crisis
* No acute leukemia in morphological relapse/persistent disease (defined as > 5% blasts in normocellular bone marrow)
* No malignant disease that is refractory to or progressive on salvage therapy
* No myelofibrosis
* Donor must be matched at HLA-A and -B at antigen level and HLA-DRB1 at allelic level

  * No available 5-6/6 HLA-A, -B, -DRB1 matched sibling donor OR 10/10 unrelated volunteer donor

PATIENT CHARACTERISTICS:

* Karnofsky performance status (PS) 60-100% OR Lansky PS 50-100% (pediatrics)
* Transaminases < 5 times upper limit of normal (ULN)
* Bilirubin < 3 times ULN
* Creatinine clearance > 50 mL/min
* DLCO > 50% predicted
* No supplemental oxygen requirements
* Not pregnant or nursing
* Negative pregnancy test
* No HIV or HTLV (I and II) antibody positivity or evidence of infection
* No acquired aplastic anemia
* No decompensated congestive heart failure or uncontrolled arrhythmia and left ventricular ejection fraction ≥ 35%
* No current active serious infection, in particular uncontrolled fungal infection
* No congenital immune deficiencies

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 6 months since prior exposure to combination chemotherapy OR only 1 course of induction combination chemotherapy for myelodysplastic syndromes or acute myeloid leukemia (please discuss with study coordinator/s if this course contained fludarabine)
* At least 6 months since prior myeloablative bone marrow transplantation
* No prior irradiation that precludes the safe administration of an additional dose of 200 cGy of total-body irradiation
* No prior autograft

Ages: 2 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-01; Primary Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Non-relapse mortality at day 100

SECONDARY OUTCOMES:
Incidence of grades II-IV and III-IV acute graft-vs-host disease (GVHD) at day 100 and chronic GVHD at 1 year
Mixed chimerism
Hemopoietic recovery

CONTACTS AND LOCATIONS:
Overall Officials: Rachael Hough, MD, Principal Investigator — University College London Hospitals
Locations (6):
- United Kingdom (6):
  - Bristol Royal Hospital for Children, Bristol, England
  - Cancer Research UK Clinical Centre at St. James's University Hospital, Leeds, England
  - University College of London Hospitals, London, England
  - UCL Cancer Institute, London, England
  - Great Ormond Street Hospital for Children, London, England
  - University of Newcastle-Upon-Tyne Northern Institute for Cancer Research, Newcastle upon Tyne, England

REFERENCES:
- [Derived] Hough R, Lopes A, Patrick P, Russell N, Raj K, Tholouli E, A Snowden J, Collin M, El-Mehidi N, Lawrie A, Clifton-Hadley L, Veys P, Craddock C, Mackinnon S, Cook G, Shaw B, Marks D. Primary graft failure, but not relapse, may be identified by early chimerism following double cord blood unit transplantation. Blood Adv. 2022 Apr 12;6(7):2414-2426. doi: 10.1182/bloodadvances.2021005106. PMID 34700343